CLINICAL TRIAL: NCT03484559
Title: The Assessment of Survival After In-hospital Cardiac Arrest for 2 Years in Tertiary Hospital
Acronym: IHCA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SİNAN YILMAZ, Assistant Professor, Aydin Adnan Menderes University
Other Study IDs: IHCA
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Cardiac Arrest
Keywords: In-hospital Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
Define the frequency and survival pattern of cardiac arrests in relation to the hospital day of event and etiology of arrest.

DETAILED DESCRIPTION:
Define the frequency and survival pattern of cardiac arrests in relation with event and etiology of arrest.

Investigators aims to evaluate the outcome of in-hospital cardiac arrests, focusing on the relationship between etiology and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Cases where the cardiac arrest team is called

Exclusion Criteria:

* Lack of data records of patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include all patients who develop in-hospital cardiac arrest. (Adnan Menderes University Training and Research Hospital).
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-05-30 (Estimated); Study Completion 2018-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of in-hospital cardiac arrest | baseline
  Incidence of in-hospital cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Sinan Yilmaz, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Adnan Menderes University Training and Research Hospital, Aydin, Turkey (Türkiye)